CLINICAL TRIAL: NCT07368023
Title: A Retrospective Study of Safety and Efficacy of Locoregional Therapies Combined With Anti-VEGF/TKIs and Immune Checkpoint Inhibitors for All Comers of Intention-to-treat Patients With Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Principal Investigator, Caide Lu, Chief Physician, Ningbo Medical Center Lihuili Hospital
Other Study IDs: KY2025PJ484
Record Dates: First submitted 2025-12-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Carcinoma Non-resectable
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initially Unresectable HCC with Conversion Therapy: This cohort consists of patients with hepatocellular carcinoma (HCC) that was initially assessed as unresectable (due to surgical inoperability or oncological unresectability per multidisciplinary team evaluation) but intended for curative treatment. All patients in this cohort received multimodal conversion therapy between January 2018 and December 2024. The therapy aimed to downstage the tumor and primarily included a combination of locoregional therapies (LRT) (such as TACE, HAIC, or radiotherapy) and systemic drug therapy (including anti-VEGF/tyrosine kinase inhibitors and immune checkpoint inhibitors). Patient data are collected retrospectively from electronic medical records and the HCC clinical database.
  Interventions: Combination Product: Locoregional Therapy (LRT) + Systemic Drug Therapy
- Initially Resectable HCC: This cohort consists of patients with hepatocellular carcinoma (HCC) that was initially assessed as resectable and suitable for curative surgery per multidisciplinary team evaluation. All patients in this cohort underwent direct radical resection (curative-intent surgery) as the primary treatment between January 2018 and December 2024, without receiving prior locoregional or systemic conversion therapy. Patient data are collected retrospectively from electronic medical records and the HCC clinical database.

INTERVENTIONS:
Combination Product: Locoregional Therapy (LRT) + Systemic Drug Therapy — Treatment regimens, doses, and durations varied based on individual clinical decisions and are collected retrospectively.
  Groups: Initially Unresectable HCC with Conversion Therapy

SUMMARY:
This is a single-center, retrospective cohort study aiming to evaluate the safety and efficacy of a combined conversion therapy strategy for patients with initially unresectable hepatocellular carcinoma (HCC).The primary objective is to assess the outcomes of intention-to-treat (ITT) patients who received multidisciplinary conversion therapy. This therapy combines locoregional treatments (LRT, such as TACE or radiotherapy) with systemic therapy (anti-VEGF/tyrosine kinase inhibitors and immune checkpoint inhibitors) with the goal of down-staging tumors to allow for subsequent curative resection.

The study plans to enroll 300 subjects. The exposure group will include approximately 100 patients with initially unresectable HCC who received the combined conversion therapy between January 2018 and December 2024. A control group of about 200 patients with initially resectable HCC who underwent direct radical surgery during the same period will be used for comparison. Data will be collected retrospectively from hospital electronic medical records and the HCC clinical database, with follow-up until December 2025.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years or older.
* Clinical and/or pathological diagnosis of hepatocellular carcinoma (HCC). China Liver Cancer (CNLC) stage I, II, or IIIA.
* Assessed by a multidisciplinary team (MDT) as having initially unresectable HCC.

Exclusion Criteria:

* Presence of extrahepatic metastasis.
* Presence of Cheng's type IV portal vein tumor thrombus (PVTT).
* Presence of Cheng's type II or III inferior vena cava tumor thrombus (IVCTT).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective single-center cohort study includes 300 HCC patients (2018-2024), divided by initial resectability:
  Initially Unresectable HCC Cohort（N=100）: Received multimodal conversion therapy (LRT + anti-VEGF/TKIs + ICIs) aiming to downstage tumors for resection.
  Initially Resectable HCC Cohort（N=200）: Underwent direct radical resection without prior conversion therapy.
  Patients were aged ≥16 with CNLC stage I-IIIA HCC. Exclusions: extrahepatic metastasis or Cheng's type IV PVTT/type II-III IVCTT. Data are collected retrospectively from EMR and an HCC database.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Conversion Rate | From the start of conversion therapy until the completion of therapy (assessed up to 24 months).
  Proportion of ITT patients with initially unresectable HCC successfully down-staged to resectability after conversion therapy (per MDT reassessment).
1-, 2-, and 3-year OS in ITT Population | Starting from conversion therapy, evaluate at 1, 2, and 3 years.
  Proportion of patients in the ITT population alive at 1, 2, and 3 years after initiation of conversion therapy (Kaplan-Meier method).
Resection Rate After Conversion | From the start of conversion therapy to the day of surgery (with a maximum evaluation period of 24 months).
  Proportion of patients who successfully undergo curative resection after down-staging.

CONTACTS AND LOCATIONS:
Overall Officials: Caide Lu, Professor, Principal Investigator — Ningbo Medical Centre Lihuili Hospital
Locations (1):
- Ningbo Medical Centre Lihuili Hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding the sharing of individual participant data (IPD) has not yet been made. The research team is currently assessing the feasibility, institutional policies, and ethical considerations related to data de-identification and sharing. A final plan will be determined prior to the completion of the study